CLINICAL TRIAL: NCT02504138
Title: A Comparison of Propofol Based Total Intravenous Anesthesia and Desflurane Based Balanced Anesthesia on Hepatic Protection During Living-donor Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2013-0454
Record Dates: First submitted 2015-07-13; First posted 2015-07-21 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane balanced anesthesia group (Experimental)
  Interventions: Drug: Desflurane balanced anesthesia
- Propofol total intravenous anesthesia group (Active Comparator)
  Interventions: Drug: Propofol total intravenous anesthesia

INTERVENTIONS:
Drug: Desflurane balanced anesthesia — Desflurane balanced anesthesia induced with thiopental sodium, remifentanil and atracurium and maintained with remifentanil target controlled infusion and desflurane inhalation
  Arms: Desflurane balanced anesthesia group
Drug: Propofol total intravenous anesthesia — Propofol total intravenous anesthesia induced with propofol, remifentanil and atracurium and maintained with remifentanil and propofol target controlled infusion
  Arms: Propofol total intravenous anesthesia group

SUMMARY:
Renal ischemia/reperfusion (I/R)-induced injury is known to be associated with immediate and long-term hepatic dysfunction after liver transplantation. Protecting the liver against I/R injury and maintaining hepatic function during transplant surgery is therefore very important in order to improve post-operative outcome. This purpose of this study is to investigate whether propofol anesthesia done in both liver donors and recipients during living-donor liver transplantation is effective in reducing liver I/R injury via its antioxidant and antiinflammatory properties and improve post-transplant outcome compared to desflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

(1) Adult liver donors and recipients scheduled for liver transplantation

Exclusion Criteria:

1. Patient refusal
2. Hypersensitivity to propofol, soybeans or peanuts
3. History of vitamin C or E intake within 5 days before surgery
4. History of acute myocardial infarct within 6 months before surgery
5. Congestive heart failure (NYHA III-IV)
6. Autoimmune disease patients
7. BMI over 30 kg/m2
8. Left ventricular ejection fraction less than 35% upon preoperative echocardiography

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
hepatic function | from 48hr before anesthesia, 1 hour after reperfusion, 1 hour after end of operation, every 24 hours daily up to 7 days postoperatively
  The difference in hepatic function of recipients between groups after liver transplantation (PT, aPTT, albumin, bilirubin, platelet count, AST, ALT, lactate, triglyceride, ammonia)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Shin S, Joo DJ, Kim MS, Bae MI, Heo E, Lee JS, Kim DW, Yoo YC. Propofol intravenous anaesthesia with desflurane compared with desflurane alone on postoperative liver function after living-donor liver transplantation: A randomised controlled trial. Eur J Anaesthesiol. 2019 Sep;36(9):656-666. doi: 10.1097/EJA.0000000000001018. PMID 31083000